CLINICAL TRIAL: NCT04440475
Title: Tap Block vs Conventional Pain Medication for Patients Undergoing Robotic Sacrocolpopexy, a Pilot Study
Brief Title: Tap Block vs Conventional Pain Medication for Patients Undergoing Robotic Sacrocolpopexy
Acronym: SACROTAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ProMedica Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 20-068
Record Dates: First submitted 2020-06-17; First posted 2020-06-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Anesthesia, Local; Prolapse; Prolapse; Female; Prolapse, Vaginal; Prolapse; Vagina, Posthysterectomy; Pain, Postoperative
MeSH Terms: conditions — Prolapse; Uterine Prolapse; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: The investigators will perform a pilot randomized control trial, where one group will be receiving TAP blocks whereas the other group will be receiving regular postoperative pain medications (acetaminophen, ibuprofen, tramadol orally upon discharge). Randomization will be completed using a computer-generated randomization sequence using 1:1 ratio with blocking in groups of 4. The randomization sequence will kept in our research office and investigators enrolling subjects will not have access. Sequentially numbered sealed opaque envelopes will be prepared following the randomization sequence, randomized participants will receive an envelope in sequential order.
  The patient and the person performing the statistical analyses will be blinded.
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient and the person performing the analysis will be masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tap Block (Experimental): TAP block at the end of the surgery, in addition to conventional postoperative oral medication as needed
  postoperative conventional oral medication as needed: Acetaminophen 650 mg Q 6 hours Ibuprofen 600 mg Q 6 hours Tramadol 50 mg Q 6 hours
  Interventions: Procedure: TAP block
- Conventional postoperative oral medication (No Intervention): postoperative conventional oral medication as needed: Acetaminophen 650 mg Q 6 hours Ibuprofen 600 mg Q 6 hours Tramadol 50 mg Q 6 hours

INTERVENTIONS:
Procedure: TAP block — Tap block description:
  The skin is prepped and draped in a sterile fashion for a lateral to posterior/lateral approach to the Transverse Abdominis Plane (TAP). The Anesthesiologists use ultrasound guidance for all TAP blocks and pre mix 60cc of 0.2% ropivicaine with 10mg of preservative free dexamethasone. After the plane is identified in approximately the mid axillary line, a 17g Tuohy needle is used under ultrasound guidance to enter the potential space from an anterior approach. The needle is visualized in-plane with the ultrasound probe, traversing the exterior and interior oblique muscles and penetrating through the posterior fascia of internal oblique into the transverse abdominal plane. Once the Tuohy is in place, the needle is aspirated and the plane is hydro-dissected using 0.2% Ropivicaine with 10mg of dexamethasone. The anesthesiologist will use 30ml of 0.2% Ropivicaine on each side.
  Arms: Tap Block

SUMMARY:
The purpose of this study is to assess whether the transversus abdominis plane block (Tap block) is different than the oral postoperative pain medications in controlling pain after robotic sacrocolpopexy.

DETAILED DESCRIPTION:
Sacrocolpopexy is a procedure to correct prolapse of the vaginal apex (top of the vagina) in women who have had a previous hysterectomy. The operation is designed to restore the vagina to its normal position and function. Pain management is an important aspect of perioperative anesthetic care. Acute postoperative pain control impacting surgical outcomes remains a controversial topic

The transversus abdominis plane (TAP) block was first presented by Rafi in 2001 as a landmark-guided technique via the triangle of Petit to achieve a field block. It involves the injection of a local anesthetic between the internal oblique muscle and transversus abdominis muscle. The thoracolumbar nerves originating from the T6 to L1 spinal roots run into this plane and supply sensory nerves to the anterolateral abdominal wall, the local anesthetic in this plane can block the neural afferents and provide analgesia to the anterolateral abdominal wall. The Tap block is a widely used procedure to help in postoperative pain management, it is easily performed, cost-effective, with minimal procedure-related morbidity. The use of Tap block is in concordance with several of the goals of Enhanced Recovery After Surgery Pathways (ERAS). In a systematic review comparing Tap bloc to no tap block for post-hysterectomy pain found that visual analog score (VAS) was lower in patients receiving tap block in both open and laparoscopic hysterectomy procedures. The study found no significant difference in the amount of morphine used by patients who underwent laparoscopic hysterectomy and received a tap block. Currently the standard of care at Promedica hospitals is to give patients oral medications to control postop pain after sacrocolpopexy. Patients are offered to receive a tap block or no, and it is up to the patient to receive the tap block or no.

No Studies on Tap block after Sacrocolpopexy have been published yet. Our hypothesis is that Tap block will reduce the need for pain meds during the first 24 to 48 hours after sacrocolpopexy.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age or older
* Planning for surgical treatment of Pelvic Organ Prolapse (POP) with robotic sacrocolpopexy and rectocele repair under general anesthesia
* Patient undergoing concurrent hysterectomy and/or sub-urethral sling will be included

Exclusion Criteria:

* Pregnant or nursing
* Allergy to ropivicaine
* History of drug/alcohol abuse
* Severe cardiovascular, hepatic, renal disease, or neurological impairment Long-acting opioid use within 3 days or any opioid use within 24 hours before surgery
* Contraindication to: acetaminophen, tramadol, non-steroidal anti- inflammatory drugs (NSAID)
* Administration of an investigational drug within 30 days before study
* Chronic pain syndromes
* Daily NSAID/opioid use
* Patients not undergoing general anesthesia
* Patients undergoing concurrent transvaginal mesh removal, anal sphincteroplasty, or fistula repair

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-06-28 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
amount of postoperative oral pain medication | 48 hours
  amount of postoperative oral pain medication used by patient after surgery
Numeric Rating Scale (NRS) scale improvement | 48 hours
  Numeric rating scale for pain will be assessed (0-10: 0 being no pain, 10 being the worst pain possible)

CONTACTS AND LOCATIONS:
Overall Officials: Dani Zoorob, MD, Principal Investigator — ProMedica Health System
Locations (1):
- Promedica Toledo Hospital, Toledo, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared with other researchers, data will be destroyed 3 years after study completion

REFERENCES:
- [Background] Yu N, Long X, Lujan-Hernandez JR, Succar J, Xin X, Wang X. Transversus abdominis-plane block versus local anesthetic wound infiltration in lower abdominal surgery: a systematic review and meta-analysis of randomized controlled trials. BMC Anesthesiol. 2014 Dec 15;14:121. doi: 10.1186/1471-2253-14-121. eCollection 2014. PMID 25580086
- [Background] Rafi AN. Abdominal field block: a new approach via the lumbar triangle. Anaesthesia. 2001 Oct;56(10):1024-6. doi: 10.1046/j.1365-2044.2001.02279-40.x. No abstract available. PMID 11576144
- [Background] Rozen WM, Tran TM, Ashton MW, Barrington MJ, Ivanusic JJ, Taylor GI. Refining the course of the thoracolumbar nerves: a new understanding of the innervation of the anterior abdominal wall. Clin Anat. 2008 May;21(4):325-33. doi: 10.1002/ca.20621. PMID 18428988
- [Background] Kim AJ, Yong RJ, Urman RD. The Role of Transversus Abdominis Plane Blocks in Enhanced Recovery After Surgery Pathways for Open and Laparoscopic Colorectal Surgery. J Laparoendosc Adv Surg Tech A. 2017 Sep;27(9):909-914. doi: 10.1089/lap.2017.0337. Epub 2017 Jul 25. PMID 28742435
- [Background] Bacal V, Rana U, McIsaac DI, Chen I. Transversus Abdominis Plane Block for Post Hysterectomy Pain: A Systematic Review and Meta-Analysis. J Minim Invasive Gynecol. 2019 Jan;26(1):40-52. doi: 10.1016/j.jmig.2018.04.020. Epub 2018 Apr 30. PMID 29723644
- [Derived] Zoorob D, Tsolakian I, Shuffle E, Perring P, Maxwell R. Addition of Transversus Abdominis Plane Block to Conventional Pain Regimens in Robotic Sacrocolpopexy Procedures-A Pilot Randomized Controlled Trial (SACROTAP). Urogynecology (Phila). 2023 Feb 1;29(2):139-143. doi: 10.1097/SPV.0000000000001287. PMID 36735426